CLINICAL TRIAL: NCT03445364
Title: Impact of Coronary Dye Injection Pressure on Myocardial Reperfusion During the Primary Percutaneous Coronary Intervention.
Brief Title: Impact of Injection Pressure on Myocardial Reperfusion During Primary PCI
Acronym: ImPress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Sestre Milosrdnice (Other)
Responsible Party: Principal Investigator, Stambuk Kresimir, M.D., Ph.D., Assisst. Prof., University Hospital Sestre Milosrdnice
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: cp0001
Record Dates: First submitted 2010-06-07; First posted 2018-02-26 (Actual); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Myocardial Reperfusion; STEMI - ST Elevation Myocardial Infarction
Keywords: Primary PCI; Coronary injection pressure; Reperfusion; Resolution of ST elevation; Myocardial Blush Grade
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low coronary injection-pressure, 200 psi (Active Comparator): Patients with STEMI who undergo Primary PCI with the use of low intracoronary dye injection pressure (of 200 psi), by using ACIST automated injector. Patients will recieve bare-metal stents at the courtasy of the interventional cardiologist, only in infarct-related artery.
  Use of different injection pressure during primary PCI
  Interventions: Other: Use of different injection pressure during primary PCI
- High coronary injection-pressure,550 psi (Active Comparator): Patients with STEMI who undergo Primary PCI with the use of higher intracoronary dye injection pressure (of 500 psi), by using ACIST automated injector. Patients will recieve bare-metal stents at the courtasy of the interventional cardiologist, only in infarct-related artery.
  Use of different injection pressure during primary PCI
  Interventions: Other: Use of different injection pressure during primary PCI

INTERVENTIONS:
Other: Use of different injection pressure during primary PCI — Using ACIST injector during the PCI it is possible to change injection pressure - in one arm low pressure of 200psi, and in the second arm average pressure of 550psi

SUMMARY:
Percutaneous coronary intervention for myocardial infarction with ST elevation could be complicated with thrombus embolisation to the more distal segments of the culprit artery. Hypothesis - lower injection pressure could reduce the incidence of this complication. In this study the investigators compare two different protocols for dye injection - first one with higher and the second one with lower injection pressure.The impact of different pressure will be evaluated using the estimation of completeness of resolution of ST elevation as well as Myocardial Blush Grade on the end of the procedure. Patents will be followed for in-hospital mortality and MACE.

DETAILED DESCRIPTION:
Distal embolization of plaque and thrombotic debris in the infarct-related artery may lead to microvascular obstruction resulting in impaired myocardial reperfusion. The aim of the study was to assess the impact of contrast injection pressure in coronary arteries, during primary percutaneous coronary intervention (PCI), on myocardial reperfusion in patients with acute ST-segment elevation myocardial infarction (STEMI).

A randomized, prospective, open label, pilot study. In the period of 6 months, consecutive patients with acute STEMI were included in the study. The acute STEMI was confirmed according to the clinical, ECG and cardioselective enzymes criteria.

Patients with the following features were eligible for inclusion: who underwent primary PCI within 12 hours from the onset of symptoms, with typical chest pain lasting >30 minutes, with ST-segment elevation of ≥1 mm in ≥2 contiguous leads in ECG and with ECGs recorded at admission, 60 minutes and 24h after primary PCI.

Exclusion criteria were: patients who had cardiogenic shock and/or underwent cardiopulmonary resuscitation before or during primary PCI, with symptoms lasting more than 12 hours, with left bundle branch block in ECG at admission, with diameter stenosis < 50% of the culprit lesion or normal coronary blood flow, with severe left main coronary artery or multivessel disease who required emergency cardiac-surgery revascularization, with permanent cardiac pacemaker or implantable cardioverter-defibrillator, with anemia (haemoglobin <100 g/L) at admission, who underwent cardiothoracic surgery or had a history of moderate or high degree valvular pathology, who had life-expectancy of less than 1 year and who did not sign informed consent. Patients were admitted through the Emergency Department, where they were evaluated for onset and duration of pain, co-morbidities and risk factors. Vital signs and complete physical status were recorded. All patients underwent 12-lead ECG and patients with acute STEMI were taken immediately to the catheterization laboratory for primary PCI.

All patients who met the inclusion criteria were randomized into two groups by means of sealed envelopes.

ELIGIBILITY:
Inclusion Criteria:

* Acute myocardial infarction with ST elevation
* Less than 12 hours of symptoms beginning
* Clear indication for primary PCI
* No contraindication for primary PCI
* Age 18 to 85

Exclusion Criteria:

* Cardiogenic or any other shock
* More than two culprit lesions/vessels
* Any major complication during PCI
* Unsuccessful intervention

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-04-01 (Actual); Primary Completion 2010-09-30 (Actual); Study Completion 2010-12-01 (Actual)

PRIMARY OUTCOMES:
Myocardial Blush Grade | At the day of inclusion in the study; at the begining og the PCI procedure and second measure - 2 minutes before the end of the primary PCI, at the last cine of the infarct related artery and the corresponding myocardium
  Myocardial Blush grade 0 to 3 (the highest)

SECONDARY OUTCOMES:
Completeness of resolution of ST segment elevation | At the first day of the inclusion in the study; ECG at admission and ECG at 60 to 90 minutes after the primary PCI procedure
  ST Segment Elevation in milimeters will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Tomislav Krcmar, M.D., Principal Investigator — University Hospital Sestre Milosrdnice
Locations (1):
- University Hospital "Sestre milosrdnice", Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No
Only complete study data of all 100 patients recruited so far, will be shared if needed

REFERENCES:
- [Derived] Stambuk K, Krcmar T, Zeljkovic I. Impact of intracoronary contrast injection pressure on reperfusion during primary percutaneous coronary intervention in acute ST-segment elevation myocardial infarction: A prospective randomized pilot study. Int J Cardiol Heart Vasc. 2019 Aug 20;24:100412. doi: 10.1016/j.ijcha.2019.100412. eCollection 2019 Sep. PMID 31463362